CLINICAL TRIAL: NCT00630201
Title: An Open-Label, Multi-Center Extension Study Of Probuphine in Patients With Opioid Dependence
Brief Title: Extension to Safety and Efficacy of Probuphine in the Treatment of Opioid Dependence
Acronym: PRO-807
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Titan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-807
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2017-06

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; opioid addiction; buprenorphine; methadone; heroin; implant; opioid withdrawal; opioid pain medication; suboxone
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Probuphine (Experimental): buprenorphine implant
  Interventions: Drug: Probuphine (buprenorphine implant)

INTERVENTIONS:
Drug: Probuphine (buprenorphine implant) — Implantable formulation of buprenorphine made of buprenorphine HCl/ethylene vinyl acetate, considered a drug. (4 implants, 6-month duration).

SUMMARY:
Buprenorphine (BPN) is an approved treatment for opioid dependence; however, in taking oral tablets, patients experience withdrawal and cravings when the variable BPN levels in the blood are low. Probuphine (buprenorphine implant) is an implant placed just beneath the skin that contains BPN. It is designed to provide 6 months of stable BPN blood levels. This study will test the safety and efficacy of Probuphine in the treatment of patient with opioid dependence. Patients who have completed 24 weeks of treatment in the Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study of Probuphine in Patients with Opioid Dependence, will be re-treated with Probuphine over an additional 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent prior to conduct of any study-related procedures
* Completed 24 weeks of treatment in PRO-805
* Deemed appropriate for entry into this extension study by the Investigator
* Females of childbearing potential and fertile males must use a reliable means of contraception

Exclusion Criteria:

* Presence of aspartate aminotransferase (AST) levels ≥ 3 X upper limit of normal and/or alanine aminotransferase (ALT) levels ≥ 3 X upper limit of normal and/or total bilirubin ≥ 1.5 X upper limit of normal and/or creatinine ≥ 1.5 X upper limit of normal
* Current diagnosis of chronic pain requiring opioids for treatment
* Pregnant or lactating females
* Current use of agents metabolized through cytochrome P450 3A4 (CYP 3A4) such as azole antifungals (e.g., ketoconazole), macrolide antibiotics (e.g., erythromycin), and protease inhibitors (e.g., ritonavir, indinavir, and saquinavir)
* Current anti-coagulant therapy (such as warfarin) or an INR > 1.2
* Current use of benzodiazepines other than physician prescribed use
* Significant medical or psychiatric symptoms, cognitive impairment, or other factors which in the opinion of the Investigator, would preclude compliance with the protocol, patient safety, adequate cooperation in the study, or obtaining informed consent
* Concurrent medical conditions (such as severe respiratory insufficiency) that may prevent the patient from safely participating in study; and/or any pending legal action that could prohibit participation and/or compliance in study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as a measure of safety | approx. 26 weeks
  Adverse events that occurred after the signing of the informed consent until 14 days after study drug treatment has been discontinued, or AEs designated as possibly-related to study drug and all Serious AEs until resolution or stabilization, were followed.

SECONDARY OUTCOMES:
Buprenorphine concentration in plasma | 24 weeks
Percent of urine samples that are negative for illicit opioids | 24 weeks
Percent of subjects retained as a measure of efficacy | 24 weeks
Percent of subjects reporting illicit drug use as a measure of efficacy | 24 weeks
Average daily dose of supplemental sublingual buprenorphine as a measure of efficacy | 24 weeks
Mean total score on SOWS as a measure of efficacy | 24 weeks
Mean total score on COWS as a measure of efficacy | 24 weeks
Mean subjective opioid cravings scores as a measure of efficacy | 24 weeks
Mean composite score Drug Problems area of Addiction Severity Index | Baseline and End of Treatment
Patient-rated Opioid use and Problems Responder Analysis as a measure of efficacy | 24 weeks
Physician-rated severity of opioid use and symptoms Responder Analysis as a measure of efficacy | 24 weeks

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Synergy Clinical Research Center, National City, California
  - Amit Vijapura, MD, Jacksonville, Florida
  - Fidelity Clinical Research, Inc., Lauderhill, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Behavioral Biology Research Unit, Johns Hopkins Bayview Campus, Baltimore, Maryland
  - Dual Diagnosis Unit, SSTAR: Stanley Street Treatment and Resources, Inc., Fall River, Massachusetts
  - Wayne State Univ. School of Medicine, Dept of Psychiatry & Behavioral Neuroscience, Detroit, Michigan
  - Psych Care Consultants Research, St Louis, Missouri
  - New York VA Medical Center, NYU School of Medicine, New York, New York
  - Duke Addictions Program, Durham, North Carolina
  - Pahl Pharmaceutical Research, LLC, Oklahoma City, Oklahoma
  - University of Pennsylvania, Treatment Research Center, Philadelphia, Pennsylvania
  - Providence Behavioral Health Services, Everett, Washington
  - Puget Sound Health CareSystem, Seattle, Washington